CLINICAL TRIAL: NCT03946176
Title: XUANRO4 - NATURE 3.2 - Nuovo Approccio Per la Riduzione Delle Tossine Uremiche Renali, REGIONE PUGLIA - FSC 2007-2013 Ricerca. Intervento "Cluster Tecnologici Regionali"
Brief Title: NATURE 3.2_New Approach for the Reduction of REnal Uremic Toxins
Acronym: NATURE32
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: XUANRO4-NATURE 3.2
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-01

CONDITIONS: Hemodialysis
Keywords: uremic toxins; gut microbiota dysbiosis; symbiotic; divinylbenzene cartridge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symbiotic (Experimental): HD patients with 7 weeks symbiotic administration + 1 week overlapping with the 3 dialytic sessions with the DVB cartridge
  Interventions: Dietary Supplement: Symbiotic; Device: DVB cartridge
- Placebo (Placebo Comparator): HD patients with 7 weeks placebo administration + 1 week overlapping with the 3 dialytic sessions with the DVB cartridge
  Interventions: Dietary Supplement: Placebo; Device: DVB cartridge

INTERVENTIONS:
Dietary Supplement: Symbiotic — HD patients follow a 8-weeks oral administration of the symbiotic supplement (2 bags/day)
  Arms: Symbiotic
Dietary Supplement: Placebo — HD patients follow a 8-weeks oral administration of the placebo (2 bags/day)
  Arms: Placebo
Device: DVB cartridge — On the last week of the symbiotic/placebo period, patients undergo 3 dialytic sessions with the DVB cartridge

SUMMARY:
The objective of the pilot study is to validate a combined approach based on the use of an innovative symbiotic and an innovative dialysis cartridge in patients on hemodialysis (HD).

The symbiotic consists of a mixture of probiotics (Lactobacilli and Bifidobacteria), prebiotics (fructoligosaccharides and inulin) and natural antioxidants (a mix of quercetin, resveratrol and proanthocyanidins).

The cartridge is composed of a divinylbenzene (DVB) adsorbing resine, expected to have high affinity to protein-bound uremic toxins pCS and IS, on the basis of its chemical structure.

This combined approach will be aimed at achieving two main objectives:

1. reduction of blood levels of microbial-derived uremic toxins, involved in cardiovascular complications
2. reduction of inflammation markers and oxidative stress and reduction of intestinal permeability

ELIGIBILITY:
Inclusion Criteria:

* CKD patients on bicarbonate hemodialysis
* Aged between 30 to 65
* BMI between 18.5 and 29.9
* Omnivore diet
* Informed consent signed

Exclusion Criteria:

* Use of antibiotics or probiotics up to 30 days prior to recruitment
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion or clinical diagnosis of malignancy
* Chronic liver disease
* Treatment with corticosteroids or immunosuppressive drugs
* Psychiatric conditions reducing the compliance to treatment protocols

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Change of serum concentration of pCS | 8 weeks
  Change of p-cresyl sulfate (pCS) serum concentrations assessed by liquid chromatography/mass spectrometry

SECONDARY OUTCOMES:
Change of serum concentration of IS | 8 weeks
  Change of indoxyl sulfate (IS) serum concentrations assessed by liquid chromatography/mass spectrometry
Change of serum concentration of D-lactate | 8 weeks
  Change of D-lactate serum concentration (uM)
Change of serum concentration of LPS | 8 weeks
  Change of lipopolysaccharide (LPS) serum concentration (EU/ml)
Change of serum concentration of inflammatory markers | 8 weeks
  Change of interleukin (IL)IL10, IL17, pentraxin3 (PTX3) serum concentrations (pg/ml) evaluated by ELISA
Change of serum concentration of NO | 8 weeks
  Change of nitric oxide (NO) serum concentration (uM) evaluated by spectrometry

OTHER OUTCOMES:
Gut microbiota | 8 weeks
  Change of the relative abundance (%) of Operational Taxonomic Units (OTUs) of Firmicutes, Bacteroidetes,Proteobacteria, Verrucomicrobia, Actinobacteria, Synergistetes, Cyanobacteria, Euryarchaeota, Chloroflexi, Nitrospirae, Tenericutes, Fusobacteria, Thermotogae, Acidobacteria evaluated by fecal bacterial DNA genome sequencing.
Change of GI symptoms | 8 weeks
  Change of gastrointestinal symptoms evaluated by Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire (15 items scored 1-7 each, 1 representing the best and 7 the worse outcome for each item)
Change of stool type | 8 weeks
  Change of stool type evaluated by BRISTOL Stool Scale (range 1-7, lower and higher values representing worse outcome, middle values representing better outcome)
Change of serum concentration of TMAO | 8 weeks
  Change of trimethylamine-N-oxide (TMAO) serum concentrations assessed by liquid chromatography/mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari
Locations (1):
- AOUConsorziale Policlinico Di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided